CLINICAL TRIAL: NCT04209348
Title: Project Wellness: A Pilot Feasibility Randomized Controlled Trial
Brief Title: The Project Wellness Pilot Feasibility Randomized Controlled Trial
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Tennessee, Knoxville (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Health Services Research
Other Study IDs: UTGSM-04547; K01DK105106 (NIH)
Record Dates: First submitted 2019-12-13; First posted 2019-12-24 (Actual); Results first posted 2024-02-12 (Actual); Last update posted 2024-02-12 (Actual); Status verified 2024-01

CONDITIONS: Diabetes, Gestational
Keywords: Exercise; Contraception; Vaccination
MeSH Terms: conditions — Diabetes, Gestational; Motor Activity

STUDY DESIGN:
Who Masked: Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Physical Activity Intervention (Experimental): The behavioral physical activity (PA) intervention focuses on walking, or stepping in place when it is not possible to walk (e.g., stormy weather). The primary goal of the PA intervention is to achieve at least 30 minutes per day of walking/stepping in place. The secondary goal is to use a PA tracker (e.g., the Fitbit Charge 3 provided by the intervention) to log and review walking/stepping, and to accumulate at least 3,000 steps during their 30 minutes of walking/stepping each day.
  Interventions: Behavioral: Physical Activity Intervention
- Wellness Education (Active Comparator): The Wellness Education intervention will deliver information on mom and baby wellness that is unrelated to physical activity, diet, metabolism, or weight (e.g., immunizations during pregnancy and encouragement to immunize the baby on schedule, postpartum contraceptive options and developing a contraceptive plan, infant car seats & safety checks).
  Interventions: Other: Wellness Education

INTERVENTIONS:
Behavioral: Physical Activity Intervention — Motivational interviewing techniques helped participants set reasonable, specific, and achievable individual goals at each session: a duration (i.e., minutes) and frequency (i.e., days of the week) of walking or stepping, and potentially, a step count (i.e., a proxy for intensity). Individual goals often differed from the program goal in an effort to meet the participants 'where they are'.
  Other Names: Step Up Program
  Arms: Physical Activity Intervention
Other: Wellness Education — The following topics were addressed: postpartum contraception, maternal immunizations, infant immunizations, car seat safety and planning for your hospital stay, and safe sleep and skin to skin. No information on PA was provided to the control group (i.e., neither encouragement for PA nor instructions to limit PA).
  Other Names: Next Steps
  Arms: Wellness Education

SUMMARY:
This pilot feasibility randomized controlled trial will be conducted among women at risk for or diagnosed with gestational diabetes (GDM) at the University of Tennessee Medical Center Knoxville (UTMC). The trial will be called Project Wellness. It will compare a physical activity (behavior change) intervention (i.e., walking/stepping in place) versus a general wellness intervention (e.g., health education focusing on immunizations, contraceptive options following delivery, etc.) on physical activity levels, maternal glycemic profile in the third trimester, and infant size and anthropometric measurements soon after birth (i.e., weight, length, circumference, skinfolds). It is hypothesized that the physical activity intervention will increase physical activity levels, and improve maternal glycemic profile and infant anthropometric measures at birth. It is also hypothesized that maternal glycemic profile in the third trimester will be associated with infant anthropometric measurements at birth.

DETAILED DESCRIPTION:
Participants will also be followed through 12 months postpartum: Maternal weight and device-based and self-reported measures of physical activity will be assessed at 3, 6, 9 and 12 months postpartum, as well as the same infant size and anthropometric measurements assessed soon after delivery.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-40 years
* Singleton viable pregnancy with low suspicion for clinically significant abnormality or aneuploidy
* Hyperglycemia after 24 weeks identified by:

One step diagnostic procedure 75-g Oral Glucose Tolerance Test (OGTT) after an overnight fast, with plasma glucose measured fasting and at 1 and 2 hrs, and any of the following plasma glucose values are met or exceeded: Fasting: 92 mg/dL (5.1 mmol/L)

1. hr: 180 mg/dL (10.0 mmol/L)
2. hr: 153 mg/dL (8.5 mmol/L)

For the Two step diagnostic procedure, only Step 1 (i.e., at risk for GDM) is required for eligibility:

Step 1: 50-g glucose screening test (non-fasting), with plasma glucose measured at 1-hr ≥130 mg/dL

Any other abnormal value on oral glucose tolerance testing associated with macrosomia

* English speaker and comfortable completing surveys in English (i.e., no translator needed)
* Planning to remain in the area for baby's first year

Exclusion Criteria:

* Previously diagnosed with diabetes (i.e., Type I or Type II diabetes) outside of pregnancy
* Contraindications to exercise (i.e., absolute contraindications according to published recommendations for exercise during pregnancy), as follows:

Hemodynamically significant heart disease, Restrictive lung disease, Incompetent cervix/cerclage, Persistent second or third trimester bleeding, Placenta previa or vasa previa after 26 weeks gestation, Premature labor during the current pregnancy, Ruptured membranes, Preeclampsia/pregnancy-induced hypertension, severe anemia

* Currently non-smoker
* Current illicit drug use
* Current use of daily medications known to alter insulin resistance and metabolic profiles (e.g., metformin, corticosteroids, anti-psychotics)
* Currently taking medication for polycystic ovarian syndrome (PCOS) (i.e., history of PCOS okay as long as she is not currently taking medication for PCOS)

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2020-08-21 (Actual); Primary Completion 2021-09-21 (Actual); Study Completion 2022-10-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Samantha F Ehrlich, PhD, Principal Investigator — Assistant Professor
Locations (1):
- The University of Tennessee Medical Center, Knoxville, Tennessee, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Ehrlich SF, Rand B, Zite NB, Fortner KB, Paudel A, Peterson C, Maples J. Exploring the relationship between regular physical activity and the 24-hour glucose cycle in gestational glucose intolerance and gestational diabetes mellitus. Am J Obstet Gynecol. 2023 Jan;228(1):100-102. doi: 10.1016/j.ajog.2022.09.004. Epub 2022 Sep 8. No abstract available. PMID 36088987

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Physical Activity Intervention | Wellness Education
Started | 10 | 10
Completed (Completed n shown here for the Physical Activity Questionnaire Data (For the Physical Activity monitor data, there one participant who delivered early and thus did not have device data at follow-up, and another participant with damaged device data at follow-up; both were in the Wellness Intervention)) | 9 | 10
Not Completed | 1 | 0
Not completed — Lost to Follow-up | 1 | 0

BASELINE CHARACTERISTICS:
Population: The trial initially launched in December 2019 but closed in March 2020 due to the COVID-19 pandemic. It re-launched in August 2020. The flow chart with eligibility and recruitment metrics is therefore presented for December 2020 through September 2021, the period unaffected by research restrictions.
Groups:
- Physical Activity Intervention: The behavioral physical activity (PA) intervention focuses on walking, or stepping in place when it is not possible to walk (e.g., stormy weather). The primary goal of the PA intervention is to achieve at least 30 minutes per day of walking/stepping in place. The secondary goal is to use a PA tracker (e.g., the Fitbit Charge 3 provided by the intervention) to log and review walking/stepping, and to accumulate at least 3,000 steps during their 30 minutes of walking/stepping each day.
  Physical Activity Intervention: Participants in both arms will wear the CGM (FDA-regulated device)
- Wellness Education: The Wellness Education intervention will deliver information on mom and baby wellness that is unrelated to physical activity, diet, metabolism, or weight (e.g., immunizations during pregnancy and encouragement to immunize the baby on schedule, postpartum contraceptive options and developing a contraceptive plan, infant car seats & safety checks).
  Wellness Education: Participants in both arms will wear the CGM (FDA-regulated device)
- Total: Total of all reporting groups
Arm/Group | Physical Activity Intervention | Wellness Education | Total
Number analyzed (Participants) | 10 | 10 | 20
Age, Continuous [Mean (Standard Deviation); unit: years] | 32.5 (4.6) | 32.5 (3.7) | 32.5 (4.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10 | 10 | 20
  Male | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 8 | 8 | 16
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 2 | 2 | 4
Region of Enrollment [Number; unit: participants]
  United States | 10 | 10 | 20

OUTCOME MEASURES:

1. Primary Outcome: Change in Self-reported Physical Activity (Assessed by Pregnancy Physical Activity Questionnaire) From Baseline to Follow-up
Description: Change in self-reported moderate to vigorous intensity walking or running activity within the sports & exercise domain, as assessed by Pregnancy Physical Activity Questionnaire (i.e., measure at follow-up study visit minus the measure at baseline study visit).
  Reference: Chasan-Taber L, Schmidt MD, Roberts DE, Hosmer D, Markenson G, Freedson PS. Development and Validation of a Pregnancy Physical Activity Questionnaire. Med Sci Sports Exerc. 2004;36(10):1750-1760.
Time Frame: approximately 6 weeks
Measure: Mean (95% Confidence Interval); unit: MET hours per week
Arm/Group | Physical Activity Intervention | Wellness Education
Number analyzed (Participants) | 9 | 9
MET hours per week | 0.22 [-0.41 to 0.84] | -0.70 [-1.31 to -0.10]

2. Primary Outcome: Change in Physical Activity Assessed by ActiGraph Monitoring Device From Baseline to Follow-up
Description: Change in minutes per day of walk/run activity, as assessed by ActiGraph monitoring device (i.e., measure at follow-up study visit minus the measure at baseline study visit).
  Reference: Hibbing PR, Lamunion SR, Kaplan AS, Crouter SE. Estimating Energy Expenditure with ActiGraph GT9X Inertial Measurement Unit. Med Sci Sports Exerc. May 2018;50(5):1093-1102.
Time Frame: approximately 6 weeks
Measure: Mean (95% Confidence Interval); unit: Minutes per day of walk/run activity
Arm/Group | Physical Activity Intervention | Wellness Education
Number analyzed (Participants) | 9 | 8
Minutes per day of walk/run activity | 0.90 [0.53 to 1.54] | -1.58 [-2.80 to -0.90]

3. Secondary Outcome: Neonatal Subscapular Skinfolds
Description: Neonatal Subscapular Skinfolds (i.e., caliper measurement to assess neonatal body composition)
Time Frame: Within 5 days of birth
Population: Subscapular skinfolds
Measure: Mean (95% Confidence Interval); unit: mm
Arm/Group | Physical Activity Intervention | Wellness Education
Number analyzed (Participants) | 7 | 10
mm | 4.37 [3.65 to 5.08] | 5.24 [4.64 to 5.84]

4. Secondary Outcome: Birthweight-for-gestational-age Z-score
Description: Birthweight-for-gestational-age Z-score based on the sex- and gestational-age-specific birth-weight distributions of the 2017 U.S. Natality files.
  Z-scores more extreme than -1.645 and +1.645 indicate birthweight-for-gestational-age-and-sex at <10th and >90th percentiles, respectively, and thus indicate increased risks for adverse health outcomes (as the relationship is U-shaped). A Z-score of 0 represents birthweight-for-gestational-age-and-sex at the 50th percentile.
  Reference: Aris IM, Kleinman KP, Belfort MB, Kaimal A, Oken E. A 2017 U.S. Reference for Singleton Birth Weight Percentiles Using Obstetric Estimates of Gestation. Pediatrics. Jul 2019;144(1).
Time Frame: Within 5 days of birth
Measure: Mean (95% Confidence Interval); unit: Z-score
Arm/Group | Physical Activity Intervention | Wellness Education
Number analyzed (Participants) | 10 | 10
Z-score | -0.87 [-1.51 to -0.24] | -0.064 [-0.70 to 0.57]

ADVERSE EVENTS:
Time Frame: Approx. 6 weeks
Description: Note that adverse events were not collected for the neonates.
Arm/Group | Physical Activity Intervention | Wellness Education
All-Cause Mortality (participants affected / at risk) | 0/10 | 0/10
Serious Adverse Events (participants affected / at risk) | 0/10 | 0/10
Other Adverse Events (participants affected / at risk) | 0/10 | 0/10

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (3):
  • Study Protocol (2020-10-26): https://cdn.clinicaltrials.gov/large-docs/48/NCT04209348/Prot_001.pdf
  • Statistical Analysis Plan (2023-08-08): https://cdn.clinicaltrials.gov/large-docs/48/NCT04209348/SAP_002.pdf
  • Informed Consent Form (2021-05-14): https://cdn.clinicaltrials.gov/large-docs/48/NCT04209348/ICF_000.pdf